CLINICAL TRIAL: NCT02726074
Title: Multicenter, Open-label Trial Evaluating the Efficacy and Safety of Perampanel Added to Monotherapy in Patients With Partial Onset Seizures With or Without Secondary Generalization
Brief Title: Trial Evaluating the Efficacy and Safety of Perampanel Added to Monotherapy in Participants With Partial Onset Seizures With or Without Secondary Generalization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-M065-412
Record Dates: First submitted 2016-03-24; First posted 2016-04-01 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2019-12

CONDITIONS: Epilepsy
Keywords: epilepsy; partial-onset seizures; secondarily generalized seizures
MeSH Terms: conditions — Epilepsy | interventions — perampanel

ARMS (1):
- Perampanel 12 mg (Experimental): During the Titration Period, participants will receive perampanel 2 milligrams per day (mg/day) and be up-titrated in no less than 2-week intervals in increments of 2 mg up to 12 mg according to the investigator's judgment. Upon entering the Maintenance Period, participants will receive the last dose they achieved at the end of the Titration Period and will continue receiving this dose once daily for the remainder of the study.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel
  Other Names: E2007

SUMMARY:
This is a multi-center, open-label, single-arm, phase 4 study to evaluate the efficacy of perampanel added to monotherapy for partial onset seizures with or without secondarily generalized seizures (total seizures).

DETAILED DESCRIPTION:
This multi-center, open-label, single-arm study evaluating the efficacy of perampanel added to monotherapy for partial onset seizures consists of 2 periods: Titration Period (12 weeks) and Maintenance Period (24 weeks). During the Titration Period, participants will begin receiving perampanel 2 milligrams per day (mg/day) and be up-titrated in no less than 2-week intervals in increments of 2 mg up to 12 mg according to the investigator's judgment. Upon entering the Maintenance Period, participants will receive the last dose they achieved at the end of the Titration Period and will continue receiving this dose once daily for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of epilepsy with partial onset seizures with or without secondarily generalized seizures according to the International League Against Epilepsy's Classification of Epileptic Seizures (1981)
* Need an initial add-on therapy after failure to control seizures with the first or further monotherapy at the optimal dose and duration
* Despite antiepileptic drug (AED) treatment within the last 8 weeks, participants must have had greater than or equal to 2 partial onset seizures, and the interval between those seizures should be more than 24 hours prior to Visit 1 (Week 0).
* Are currently being treated with stable doses of monotherapy for 8 weeks prior to Visit 1 (Week 0) (Standard AEDs)
* If antidepressants or antianxiety drugs are used, participants must be receiving stable doses and administrations of antidepressants or antianxiety drugs for 8 weeks prior to Visit 1 (Week 0)

Exclusion Criteria:

* Females who are pregnant (positive beta-human chorionic gonadotropin (β-hCG test) or breastfeeding
* Presence of previous history of Lennox-Gastaut syndrome
* Presence of nonmotor simple partial seizures only
* Presence of primary generalized epilepsies or seizures such as absences and/or myoclonic epilepsies
* A history of status epilepticus within 12 weeks before Visit 1 (Week 0)
* Participants on antipsychotics or who have psychotic disorder(s) or unstable recurrent affective disorder(s) with a history of attempted suicide within 1 year before Visit 1 (Week 0)
* Presence of a progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors
* Concomitant use of barbiturates (except for seizure control indication and premedication for electroencephalogram [EEG]) and benzodiazepines (except for seizure control indication) within 8 weeks prior to Visit 1 (Week 0)
* Use of intermittent rescue benzodiazepines (that is, 1 to 2 doses over a 24-hr period considered one-time rescue) 2 or more times in an 8-week period prior to Visit 1 (Week 0)
* Participant who is participating in other intervention clinical trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Busan
  - Daegu
  - Daejeon
  - Gwangju
  - Seongnam
  - Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 11 investigative sites in Korea from 03 May 2016 to 26 April 2018.
Pre-assignment Details: A total of 106 participants were enrolled in this study, 102 participants were included in the safety set excluding 3 participants who did not received the investigational product and 1 participant who was not assessed for safety at least once after study treatment.
Groups:
- Perampanel 12 mg: During the Titration Period, participants received perampanel 2 milligrams per day (mg/day) and were up-titrated in no less than 2-week intervals in increments of 2 mg up to 12 mg according to the investigator's judgment. Upon entering the Maintenance Period, participants received the last dose they achieved at the end of the Titration Period and continued receiving this dose once daily for up to Week 36. At the discretion of investigators, dose adjustments were allowed based on the participant's clinical response and tolerability.
Period: Overall Study
Arm/Group | Perampanel 12 mg
Started | 106
Treated | 102
Completed | 80
Not Completed | 26
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 14
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 2
Not completed — Others | 3

BASELINE CHARACTERISTICS:
Population: The full analysis set included participants who received at least one dose of investigational product and were assessed for primary efficacy at least once after study treatment.
Groups:
- Perampanel 12 mg: During the Titration Period, participants received perampanel 2 mg/day and were up-titrated in no less than 2-week intervals in increments of 2 mg up to 12 mg according to the investigator's judgment. Upon entering the Maintenance Period, participants received the last dose they achieved at the end of the Titration Period and continued receiving this dose once daily for up to Week 36. At the discretion of investigators, dose adjustments were allowed based on the participant's clinical response and tolerability.
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.25 (14.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: 50 Percent (%) Responder Rate for Partial Onset Seizure With or Without Secondary Generalization
Description: The 50% responder rate was defined as the percentage of participants who achieved at least 50% reduction from baseline in the frequency of partial onset seizure with or without secondary generalization during the Maintenance Period.
Time Frame: Baseline up to Week 36
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 85
percentage of participants | 80.0 [69.92 to 87.90]

2. Secondary Outcome: 75% Responder Rate for Partial Onset Seizure With or Without Secondary Generalization
Description: The 75% responder rate was defined as the percentage of participants who achieved at least 75% reduction from baseline in the frequency of partial onset seizure with or without secondary generalization during the Maintenance Period.
Time Frame: Baseline up to Week 36
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 85
percentage of participants | 71.76 [60.96 to 81.00]

3. Secondary Outcome: 100% Responder Rate (Seizure Free Rate) for Partial Onset Seizure With or Without Secondary Generalization
Description: The 100% responder rate was defined as the percentage of participants who achieved at least 100% reduction from baseline in the frequency of partial onset seizure with or without secondary generalization during the Maintenance Period.
Time Frame: Baseline up to Week 36
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 85
percentage of participants | 47.06 [36.13 to 58.19]

4. Secondary Outcome: Percent Change From Baseline in Partial Onset Seizure Frequency With or Without Secondary Generalization to the Titration and Maintenance Period
Description: Percent change in the frequency of partial onset seizure with or without secondary generalization was defined as the percent reduction in seizure frequency from baseline to titration period and maintenance period. Percent change from Baseline was calculated as: ([post-Baseline value minus the Baseline value] / Baseline value)*100. A negative percent change from baseline indicates a decrease in partial seizure frequency.
Time Frame: Weeks 12 and 36
Population: The full analysis set included participants who received at least one dose of investigational product and were assessed for primary efficacy at least once after study treatment. Participants who were evaluable for this given measure at a given time point were included for this assessment.
Measure: Median (Full Range); unit: percent change
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 85
percent change
  Percent Change at Week 12 | -90.48 [-100.00 to 317.25]
  Percent Change at Week 36: number analyzed (Participants) | 84
  Percent Change at Week 36 | -95.02 [-100.00 to 1457.33]

5. Secondary Outcome: 50% Responder Rate in Secondary Generalized Tonic Clonic (GTC) Seizures
Description: The 50% responder rate was defined as the percentage of participants who have achieved at least a 50% reduction from baseline in the frequency of secondary GTC seizure during the Maintenance Period. GTC seizures are defined as seizures involved with generalized stiffening and rhythmic jerking of the limbs, caused by bilateral malfunction of the brain.
Time Frame: Baseline up to Week 36
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 16
percentage of participants | 87.50 [61.65 to 98.45]

6. Secondary Outcome: 75% Responder Rate in Secondary GTC Seizures
Description: The 75% responder rate was defined as the percentage of participants who achieved at least a 75% reduction from baseline in seizure frequency of secondary GTC seizure during the Maintenance Period. GTC seizures are defined as seizures involved with generalized stiffening and rhythmic jerking of the limbs, caused by bilateral malfunction of the brain.
Time Frame: Baseline up to Week 36
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 16
percentage of participants | 87.50 [61.65 to 98.45]

7. Secondary Outcome: 100% Responder Rate (Seizure Free Rate) in Secondary GTC Seizures
Description: The 100% responder rate was defined as the percentage of participants who have at least a 100% reduction from baseline in the frequency of secondary GTC seizures during the Maintenance Period. GTC seizures are defined as seizures involved with generalized stiffening and rhythmic jerking of the limbs, caused by bilateral malfunction of the brain.
Time Frame: Baseline up to Week 36
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 16
percentage of participants | 75.00 [47.62 to 92.73]

8. Secondary Outcome: Percent Change From Baseline in Secondary GTC Seizure Frequency to the Titration and Maintenance Period
Description: Percent change in the frequency of secondary GTC seizure was defined as the percent reduction in seizure frequency from baseline to Titration Period and Maintenance Period. GTC seizures are defined as seizures involved with generalized stiffening and rhythmic jerking of the limbs, caused by bilateral malfunction of the brain. Percent change from Baseline was calculated as: ([post-Baseline value minus the Baseline value] / Baseline value)*100. A negative percent change from baseline indicates a decrease in partial seizure frequency.
Time Frame: Weeks 12 and 36
Population: as for outcome 4
Measure: Median (Full Range); unit: percent change
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 85
percent change
  Percent Change at Week 12: number analyzed (Participants) | 16
  Percent Change at Week 12 | -100.00 [-100.00 to 6.33]
  Percent Change at Week 36: number analyzed (Participants) | 15
  Percent Change at Week 36 | -100.00 [-100.00 to -19.54]

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From the first dose of investigational product to the last visit or 28 days after the last dose (up to 1 year 11 months)
Population: The safety set included participants who received at least one dose of investigational product and were assessed for safety at least once after study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Perampanel 12 mg
Number analyzed (Participants) | 102
Participants
  TEAEs | 77
  SAEs | 8

ADVERSE EVENTS:
Time Frame: From the first dose of investigational product to the last visit or 28 days after the last dose (up to 1 year 11 months)
Arm/Group | Perampanel 12 mg
All-Cause Mortality (participants affected / at risk) | 0/102
Serious Adverse Events (participants affected / at risk) | 8/102
Other Adverse Events (participants affected / at risk) | 74/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel 12 mg (N=102)
Seizure (Nervous system disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Perforation (General disorders) | 1
Furuncle (Infections and infestations) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel 12 mg (N=102)
Dizziness (Nervous system disorders) | 51
Somnolence (Nervous system disorders) | 10
Headache (Nervous system disorders) | 9
Dysarthria (Nervous system disorders) | 5
Memory impairment (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Parkinsonism (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anger (Psychiatric disorders) | 2
Irritability (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Tearfulness (Psychiatric disorders) | 1
Fatigue (General disorders) | 2
Oedema (General disorders) | 2
Face oedema (General disorders) | 1
Gait disturbance (General disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Lip injury (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Diplopia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Bicytopenia (Blood and lymphatic system disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Weight increased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Labile hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT02726074/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT02726074/SAP_001.pdf